CLINICAL TRIAL: NCT01057264
Title: A Phase I Study of Hepatic Arterial Infusion (HAI) of Abraxane in Combination With Gemcitabine and Bevacizumab for Patients With Advanced Cancers Metastatic to the Liver
Brief Title: HAI Abraxane With Gemcitabine and Bevacizumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0741; NCI-2011-00555 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-01-25; First posted 2010-01-27 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Advanced Cancers
Keywords: Liver; Cancer; Hepatic arterial infusion; HAI; Abraxane; Nab-Paclitaxel; Paclitaxel; ABI-007; Gemcitabine; Gemcitabine Hydrochloride; Gemzar; Bevacizumab; Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF; Filgrastim; G-CSF; Neupogen
MeSH Terms: conditions — Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Taxes; Albumin-Bound Paclitaxel; Gemcitabine; Bevacizumab; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HAI Abraxane + Gemcitabine + Bevacizumab (Experimental): HAI (hepatic arterial infusions) Abraxane with Gemcitabine + Bevacizumab
  Interventions: Drug: HAI Abraxane; Drug: Gemcitabine; Drug: Bevacizumab; Drug: Filgrastim

INTERVENTIONS:
Drug: HAI Abraxane — Starting dose: 120 mg/m^2 by HAI infusion over 24 hours on Day 1 of 21 day cycle
  Other Names: Nab-paclitaxel; Paclitaxel (protein bound); ABI-007
Drug: Gemcitabine — Starting dose: 600 mg/m^2 by IV on Days 1 and 8 of 21 day cycle
  Other Names: Gemzar; Gemcitabine Hydrochloride
Drug: Bevacizumab — 10 mg/kg IV on Day 1 of 21 day cycle
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Filgrastim — 5 mcg/kg subcutaneously starting at least 24 hours after Day 1 completion of chemotherapy, for 3 days.
  Other Names: G-CSF; Neupogen

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of Abraxane® (nab-paclitaxel) when given directly into the liver, in combination with Gemzar® (gemcitabine) and Avastin® (bevacizumab) when given by vein.

DETAILED DESCRIPTION:
The Study Drugs:

Nab-paclitaxel is designed to block cancer cells from dividing, which may cause the cancer cells to die.

Gemcitabine is designed to disrupt the growth of cancer cells, which may cause cancer cells to die.

Bevacizumab is designed to block the growth of blood vessels that supply the nutrients needed for tumor growth, which may prevent or slow down the growth of cancer cells. Bevacizumab is no longer FDA approved to treat breast cancer.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of the combination of nab-paclitaxel and gemcitabine based on when you join this study. Up to 6 dose levels of nab-paclitaxel and gemcitabine will be tested. All participants will receive the same dose level of bevacizumab, regardless of when you join the study. Between 3-6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level of the combination of nab-paclitaxel and gemcitabine in combination with bevacizumab. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of the combination of nab-paclitaxel and gemcitabine given in combination with bevacizumab is found.

Once the highest tolerable dose is found, up to 12 additional participants receive this dose. This is called the expansion group.

Catheter Placement:

On Day 1 of each 21-day study cycle, a catheter (a sterile, flexible tube) will be placed into a large artery that carries blood to the liver in your groin area, on the right side of the body. The area where the catheter will be placed will first be numbed with local anesthetic. The catheter will be taped in place to prevent it from moving or coming out while you are receiving nab-paclitaxel. You will lie flat on your back while receiving the study drug, and you will be on bedrest until the catheter is removed.

The doctor who performs the catheter placement procedure will explain it to you in more detail, and you will be asked to sign a separate consent form that describes the catheter placement procedure and its risks in more detail.

After the catheter is in place, you will receive heparin, a drug that is used to help prevent blood clots. Heparin will be started as soon as the catheter is placed and will continue for up to 2 hours.

The catheter will be removed right after you receive nab-paclitaxel. While the catheter is being removed, the study staff will apply pressure to your groin area for 15 minutes in order to stop the bleeding. The catheter will be in place for about 1 hour, or until the nab-paclitaxel administration is complete.

Study Drug Administration:

Nab-paclitaxel will be given through the catheter into the artery that carries blood to your liver nonstop for 1 hour starting on Day 1 of each cycle. If the study doctor thinks it is needed, you will be given drugs by vein to lower the risk of nausea before each dose as part of your standard, routine care.

Gemcitabine will be given by vein over 1 hour on Days 1 and 8 of each cycle.

Bevacizumab will be given by vein on Day 1 of each cycle. The first time you receive bevacizumab, it will be given over 90 minutes. If you tolerate it well, the rest of the doses will be given over 30-60 minutes.

If you do not tolerate the study drug combination well, the doses that you receive may be lowered. If you experience certain side effects, the study drug doses may be delayed and that study cycle may last longer than 21 days.

Starting at least 24 hours after the you receive the study drug on Day 1, you will receive Neupogen® (filgrastim) through a needle injected under the skin. You will continue to receive filgrastim for 3 days (Days 2-4). Filgrastim is being given to help prevent possible side effects related to the other study drugs.

Study Visits:

You will stay in the hospital for up to 7 days (Days 1-7 of each cycle) at the beginning of each cycle, until you recover from any side effects that you may experience. You will be seen by a doctor or "advanced practice" nurse every day while you are in the hospital to check on how you are recovering.

On Day 1 of each cycle:

* You will have a physical exam, including measurement of your weight and vital signs.
* Blood (about 3 teaspoons) will be drawn for routine tests, to test your blood's ability to clot, and tumor marker testing.

On Day 2 of each cycle:

-You will have a physical exam, including measurement of your weight and vital signs.

Every 2 cycles, or at any time the study doctor thinks it is needed, women who are able to become pregnant will have a urine pregnancy test. To remain on this study, the pregnancy test must be negative.

At the end of every 2 cycles (Cycles 2, 4, 6, and so on), or at any time the study doctor thinks it is needed, a chest x-ray, CT scan, MRI scan, PET scan and/or PET/CT scan will be performed to check the status of the disease. After 10 cycles of study drug treatment, you may have scans every 3 cycles instead of 2 cycles, if your doctor feels that this is in your best interest. If the study doctor thinks it is better for you, other types of scans that have not been listed here may be performed.

Follow-Up Visit:

Six (6) weeks after the last dose of the study drug combination, or if you stop taking the study drug combination for any reason, the following tests and procedures will be performed:

* You will have a physical exam.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) will be drawn for routine tests and to test your blood's ability to clot.
* If the study doctor thinks it is needed, a chest x-ray, CT scan, MRI scan, PET scan and/or PET/CT scan will be performed to check the status of the disease. If the study doctor thinks it is better for you, other types of scans that have not been listed here may be performed.

Length of Study:

You may continue taking the study drug combination for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse or intolerable side effects occur.

This is an investigational study. Nab-paclitaxel is FDA approved and commercially available when given by vein for the treatment of breast cancer.

Gemcitabine is FDA approved and commercially available for the treatment of pancreatic cancer, breast cancer that is metastatic (has spread to other parts of the body), non-small cell lung cancer (NSCL), and ovarian cancer. Bevacizumab is FDA approved and commercially available for the treatment of metastatic colorectal cancer, NSCL, and a type of brain cancer called glioblastoma multiforme.

Giving nab-paclitaxel into an artery that carries blood directly into the liver is investigational. Using the study drug combination for treating advanced cancer that has spread to the liver is investigational.

Up to 80 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed cancer with metastatic liver metastases.
2. Patients should be refractory to standard therapy, relapsed after standard therapy, or have no standard therapy that increases survival by at least 3 months, unless the drugs in the protocol regimen are part of the standard of care.
3. Performance status Eastern Cooperative Oncology Group (ECOG) 0-2 (capable of all self care but unable to carry out any work activities).
4. Adequate renal function (serum creatinine </= 2.0 mg/dL or the calculated glomerular filtration rate (GFR) >/= 40 mL/min if creatinine > 2.0 mg/dL).
5. Hepatic function: Total bilirubin </= 5 mg/dL, alanine transaminase (ALT) </= 5 times upper normal reference value.
6. Adequate bone marrow function (absolute neutrophil count (ANC) >/= 1500 cells/uL; platelets (PLT) >/= 100,000 cells/uL).
7. At least three weeks from previous cytotoxic chemotherapy before day 1 of hepatic arterial infusion (HAI) infusion. After targeted or biologic therapy there should be 5 half-lives or three weeks, whichever is shorter.
8. All females in childbearing age MUST have a negative urine human chorionic gonadotropin (HCG) test unless prior hysterectomy or menopause (defined as age above 55 and six months without menstrual activity). Patients should not become pregnant or breast-feed while on this study. Sexually active patients should use effective birth control.
9. Must be >/= 18 years of age.

Exclusion Criteria:

1. Pregnant females.
2. Inability to complete informed consent process and adhere to protocol treatment plan and follow-up requirements.
3. Serious or non-healing wound, ulcer or bone fracture.
4. History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days.
5. Uncontrolled systemic vascular hypertension (systolic blood pressure > 140 mm Hg, diastolic blood pressure > 90 mm Hg).
6. Uncontrolled intercurrent illness, including, but not limited to, ongoing or active infection requiring parental antibiotics, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Patients already in uncompensated liver failure (i.e. Child Pugh Liver Classification C).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Escalating Doses of Hepatic Arterial Infusions of Abraxane in Combination with Gemcitabine and Bevacizumab | 21 days
  If not more than 33% of the patients in the cohort develop dose limiting toxicities (DLT), this cohort considered maximum tolerated dose (MTD). Dose-limiting toxicity (DLT) defined as any grade 3 or 4 non-hematologic toxicity as defined in the most current version of NCI Common Toxicity Criteria for Adverse Effects (CTCAE). MTD defined by DLTs that occur in the first cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Apostolia M. Tsimberidou, MD, PHD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org